CLINICAL TRIAL: NCT00376103
Title: A Phase I/II Trial of Maximal Resection, Local Radiation Boost With Concomitant Temozolomide, Followed by External Radiation Therapy With Concomitant Temozolomide for the Treatment of Newly Diagnosed Glioblastoma Multiforme
Brief Title: Radiation Boost for Newly Diagnosed Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Loss of funding from sponsor
Sponsor: Methodist Healthcare (Other)
Responsible Party: Allen Sills, MD, Methodist Healthcare
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHIRB 2006-032
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Glioblastoma Multiforme
Keywords: Brain Tumor; GBM; Glioblastoma Multiforme; Glioblastoma; Brachytherapy; Temozolomide; Temodar
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Temozolomide; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: temozolomide — 75 mg/m2/day
  Other Names: Temodar
Procedure: Brachytherapy — 60 Gy to 1 cm
Procedure: External Beam Radiation Therapy — 60 Gy

SUMMARY:
The purpose of this study is to determine treatment related toxicity, tumor response, progression-free survival and quality of life of newly diagnosed Glioblastoma Multiforme (GBM) patients undergoing a combination of surgical resection, brachytherapy and external beam radiation with concomitant temozolomide, followed by adjuvant temozolomide.

DETAILED DESCRIPTION:
The study design is multi-centered and non-randomized. Patients with newly diagnosed GBM undergoing initial surgical resection will be candidates for this study. Eligible patients will undergo surgical resection within 30 days of diagnosis.

Newly diagnosed patients with presumed diagnosis of GBM will undergo surgery for maximal resection. After frozen section diagnosis of GBM is confirmed, the GliaSite® will be placed into the tumor cavity.

After the patient recovers from surgery, radiation therapy (60 Gy to 1 cm) is delivered via the GliaSite®. Radiation therapy with the GliaSite® will be initiated within 21 days after surgery. Concomitant temozolomide (75 mg/m2/d) is started 2 days prior to radiation therapy with the GliaSite® and continued for a total of 7 days.

Within 21 days following radiation therapy with the GliaSite®, external beam radiation therapy (60 Gy in 30 fractions) will be initiated. Concomitant temozolomide (75 mg/m2/d) will start on day 1 of external beam radiation therapy and continue through the external beam radiation therapy interval, ending with the last day of radiation.

Four weeks (+/- 2 days) after completion of external beam radiation therapy, temozolomide (150 mg/m2/d) for 5 days every 28 days will be initiated for one cycle.

At the start of cycle 2, the dose will be escalated to 200 mg/m2/d, if the CTC non-hematological toxicity for cycle 1 is Grade < 2 (except for alopecia, nausea and vomiting).

This will continue for up to a total of 12 cycles, unless disease progression or severe myelosuppression is noted.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, unifocal, unilateral, supratentorial lesion seen on MRI and suspicious for Glioblastoma Multiforme
* Subject must be a candidate for surgical resection of the tumor mass with feasible gross total resection
* Age 18 years or older
* Subject must be an appropriate candidate to receive brachytherapy and temozolomide per the GliaSite RTS and temozolomide IFU
* The tumor must be histopathologically confirmed by intra-operative frozen section and by final pathology
* Karnofsky Performance Status (KPS) => 70
* Negative pregnancy test if a female of childbearing age and not surgically sterilized
* Male or female subject agrees to use acceptable birth control methods while receiving treatment (if not surgically sterile)
* Life expectancy > 3 months
* Adequate laboratory results: ANC => 1.5 x 109/L. Platelets => 100 x 109/L
* Subject or legal representative must provide informed consent and HIPAA authorization prior to surgery

Exclusion Criteria:

* Prior use of temozolomide
* Presence or history of severe hepatic or renal impairment
* Subject cannot tolerate temozolomide therapy due to NPO status or intractable nausea and vomiting
* Subject with prior intracranial malignancy
* Major medical illness or psychiatric impairments that in the investigators opinion will prevent administration or completion of the protocol therapy
* Subject has pacemaker or other MRI non-compatible metal in the body
* Previous radiation to the head/neck or brain
* Pregnant or lactating women
* Patient has allergy to iodine and/or dacarbazine
* Creatinine > 1.5x upper limits of normal (ULN), AST > 3x ULN
* Chemotherapy within the last 6 months
* Residual tumor >1 cm (in a single dimension) on baseline MRI scan (T1 post-gadolinium images)
* Balloon surface within 1 cm of critical structure (brain stem, midbrain, optic chiasm) on baseline MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Treatment-related toxicity. | 1 year

SECONDARY OUTCOMES:
6 month, 1 year and overall survival. | End of study
Tumor progression. | End of study
Progression-free survival. | End of study
Quality of life. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Allen K Sills, MD, Principal Investigator — Methodist University Hospital
Locations (1):
- Methodist University Hospital, Memphis, Tennessee, United States